CLINICAL TRIAL: NCT00002157
Title: Compassionate Use Study of Two Dose Levels of Thalidomide in Adults With HIV Wasting Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 230B; W-002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-12

CONDITIONS: HIV Infections; HIV Wasting Syndrome
Keywords: Acquired Immunodeficiency Syndrome; Cachexia; Thalidomide
MeSH Terms: conditions — HIV Infections; HIV Wasting Syndrome; Acquired Immunodeficiency Syndrome; Cachexia | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
To allow patients with HIV-associated wasting to receive thalidomide treatment at 1 of 2 doses. To gain safety and efficacy data from a broader base of patients with HIV-associated wasting in order to support Celgene's pivotal placebo-controlled study.

DETAILED DESCRIPTION:
Patients are randomized to receive thalidomide at 1 of 2 doses for 12 weeks initially, with response assessed at weeks 2, 4, 8, and 12. Patients failing the low dose will be eligible to increase the dose to the higher dose. Treatment may continue indefinitely. After 12 weeks, patients continuing treatment are evaluated every 2 months for up to 6 additional months, then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy.
* Prophylaxis or treatment for opportunistic infection.

Patients must have:

HIV-associated wasting.

Prior Medication:

Allowed:

* Prior enrollment on Celgene's placebo-controlled thalidomide study, provided patient meets specified criteria for not continuing on that study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Celgene Corp, Warren Township, New Jersey, United States